CLINICAL TRIAL: NCT01993056
Title: The Influence of 11+ on Injury Incidence and FMS-Score in Veteran Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Collaborators: FIFA-Medical Assessment and Research Centre (F-MARC), Zurich, Switzerland (Unknown)
Responsible Party: Principal Investigator, Anne Krieg M.D., Dr, Universität des Saarlandes
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Saarland University 10/2011
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Injury
Keywords: injury incidence, male veteran soccer, 11+, Functional Movement Screen, FMS, warm-up
MeSH Terms: conditions — Wounds and Injuries

ARMS (2):
- warm-up with 11+ (Experimental): The "FIFA 11+" is a complete warm up program aiming on reduce common soccer injuries
  Interventions: Behavioral: "FIFA 11+"
- control (Placebo Comparator): the control group follows its regular training routine
  Interventions: Behavioral: no "FIFA 11+"

INTERVENTIONS:
Behavioral: "FIFA 11+"
  Arms: warm-up with 11+
Behavioral: no "FIFA 11+"
  Arms: control

SUMMARY:
According to available data the injury rate in male veteran soccer is high. Interventions to prevent injuries are requested. The 11+ warm-up program was developed by FIFA-experts and consists of several exercises with an overall-length of about 20 min. This study shall investigate the influence of 11+ on injury incidence and Functional Movement Screen (FMS)-Score in male veteran soccer players. Additionally it is to be examined if there is a relationship between FMS-Score and injury incidence. For this purpose the 11+-program is accomplished under supervised conditions over one regular season in a randomized-controlled study design. Injuries are documented via questionnaires in accordance with the FIFA-consensus-statement. FMS-Score is evaluated before and after the interventional period.

ELIGIBILITY:
Inclusion Criteria:

* male veteran soccer players aged 32 and older, who are member of a club veteran team; training and matches on a regular basis

Exclusion Criteria:

* major time-loss injury, chronic inflammatory joint disease

Min Age: 32 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
injury incidence | August 2011 - June 2012
  injury incidence (injuries per 1000h of soccer)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hammes, Principal Investigator — Saarland University, Institute for Sports and Preventive Medicine
Locations (1):
- Saarland University, Saarbrücken, Saarland, Germany